CLINICAL TRIAL: NCT03628560
Title: Alternate Methodology of Pulse Oximeter Validation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending equipment repair
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00100105
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Hypoxemia; Desaturation of Blood
Keywords: Healthy volunteer; Oximetry; Pulse oximeter; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- RespirAct Step-Wise Normocapnia desaturation sequence (Experimental): Reduction in oxygen saturation 100 to 70% in approximate 5% steps.
  Interventions: Device: RespirAct Step-Wise Normocapnia desaturation sequence
- RespirAct Slope Normocapnia desaturation sequence (Experimental): Reduction in oxygen saturation 100 to 70% as gradual slope.
  Interventions: Device: RespirAct Slope Normocapnia desaturation sequence
- RespirAct Step-Wise Hypocapnia desaturation sequence (Experimental): Reduction in oxygen saturation 100 to 70% in approximate 5% steps.
  Interventions: Device: RespirAct Step-Wise Hypocapnia desaturation sequence
- RespirAct Slope Hypocapnia desaturation sequence (Experimental): Reduction in oxygen saturation 100 to 70% as gradual slope.
  Interventions: Device: RespirAct Slope Hypocapnia desaturation sequence
- ROBD Step-Wise desaturation sequence (Active Comparator): ROBD = Reduced Oxygen Breathing Device. Reduction in oxygen saturation 100 to 70% in approximate 5% steps. This represents the standard type of desaturation sequence for pulse oximeter accuracy testing.
  Interventions: Device: ROBD Step-Wise desaturation sequence

INTERVENTIONS:
Device: RespirAct Step-Wise Normocapnia desaturation sequence — Blood carbon dioxide controlled at normal value (normocapnia).
  Arms: RespirAct Step-Wise Normocapnia desaturation sequence
Device: RespirAct Slope Normocapnia desaturation sequence — Blood carbon dioxide controlled at normal value (normocapnia).
  Arms: RespirAct Slope Normocapnia desaturation sequence
Device: RespirAct Step-Wise Hypocapnia desaturation sequence — Blood carbon dioxide controlled at lower than normal value (hypocapnia).
  Arms: RespirAct Step-Wise Hypocapnia desaturation sequence
Device: RespirAct Slope Hypocapnia desaturation sequence — Blood carbon dioxide controlled at lower than normal value (hypocapnia).
  Arms: RespirAct Slope Hypocapnia desaturation sequence
Device: ROBD Step-Wise desaturation sequence — Blood carbon dioxide is controlled at normal or lower value by subject's own breathing rate.
  Arms: ROBD Step-Wise desaturation sequence

SUMMARY:
This study will determine if the replacement of the measured arterial blood oxygen saturation with expired (end-tidal) oxygen value is an acceptable method to calculate the accuracy of pulse oximeters.

DETAILED DESCRIPTION:
Pulse oximeters are non-invasive devices that use light to display an estimate (denoted by SpO2) of the true arterial blood oxygen saturation (SaO2). The accuracy of the pulse oximeter is determined from desaturation sequences (reduction in SpO2 from 100 to 70%) performed in healthy volunteers. The current standard desaturation sequence is a step-wise reduction in 5% SpO2 increments, achieved by reduction in inspired oxygen delivered by a gas blender such as the ROBD (Reduced Oxygen Breathing Device). This mixes oxygen and nitrogen (components of air) to produce the desired gas mixture. Throughout the desaturation sequence arterial blood gas samples are drawn at each step. The blood gas samples are processed through a co-oximeter to measure the SaO2. For each SaO2 measurement there will be a corresponding SpO2 recorded. All data points from all subjects are amalgamated together to allow calculation of how well SpO2 corresponds to the SaO2 throughout the range of 70 - 100% oxygen saturation. Accuracy, A[RMS], is the unit of measure and this incorporates both bias and precision.

When the ROBD is used in a desaturation sequence, the subjects' arterial blood carbon dioxide (CO2) level will initially be normal (normocapnia). With the reduction in SpO2 during the desaturation sequence, the subjects' breathing rate will increase and this will cause the a physiological reduction in the blood CO2 value (hypocapnia). The extent of hypocapnia will vary from one subject to another. It is not known whether the presence of hypocapnia may have an effect upon the accuracy measurement.

The RespirAct is a gas blender which, in contrast to the ROBD, can control both the oxygen level as well as the carbon dioxide level. The end-tidal oxygen level (PAO2) is continuously displayed by the RespirAct during the desaturation sequence. The PAO2 closely approximates to arterial blood oxygen (PaO2) - the degree of closeness will be measured in the study. Through an accepted formula, the SaO2 can be derived from the measured PAO2. The derived SaO2 values can subsequently be used to measure the accuracy of the pulse oximeter. This A[RMS] can then be compared with the A[RMS] calculated from the blood gas co-oximeter PaO2 / SaO2 values. If the accuracies are comparable then this would remove the need for arterial line placement during pulse oximeter validation studies.

Eligible healthy volunteers will complete five (5) oxygen desaturation sequences with adjustment of sequence type and/or CO2 level. Two sequences will be delivered by step-wise reduction and two will be delivered by gradual slope. Two sequences will be delivered at normocapnia and two will be delivered at hypocapnia values. The ROBD sequence will be a step-wise reduction with CO2 value set by the subjects' own breathing control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 50 years
* Subject is willing to provide written informed consent and is able to comply with anticipated study procedures

Exclusion Criteria:

* Body Mass Index (BMI) < 18.0 or > 30.0
* Known significant respiratory, cardiovascular or medical condition that precludes study participation as judged by investigator
* Anemia [hemoglobin value below lower range of normal for gender]
* Abnormal hemoglobin electrophoresis result
* Exposure to nicotine [positive test at screening or study day]
* Abnormal drug screen [positive test at screening or on day of study]
* Positive pregnancy test for females [serum test at screening; urine test on study day]
* Abnormal Allen's test for collateral circulation
* Abnormal Electrocardiogram
* Abnormal Pulmonary Function Test
* Abnormal venous blood gas result
* Intolerance of facemask

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of FDA-approved pulse oximeter when calculated with RespirAct-derived end-tidal PAO2 values and with co-oximeter measured arterial PaO2 values | 1 study day
  The unit of measure of accuracy is called A[RMS] and is a composite value of bias and precision.
PAO2 values | 1 study day
  RespirAct-derived end-tidal PAO2 values with co-oximeter measured arterial PaO2 values

SECONDARY OUTCOMES:
Accuracy, A[RMS], when a step-wise desaturation sequence is used against a slope desaturation sequence. | 1 study day
  The unit of measure of accuracy is called ARMS and is a composite value of bias and precision.
Level of PaCO2 (hypocapnia versus normocapnia) | 1 study day

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, FRCA, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Human Pharmacology & Physiology Lab at Duke University — https://anesthesiology.duke.edu/?page_id=845005